CLINICAL TRIAL: NCT00375349
Title: Non Alcoholic Fatty Liver Disease Influence of Statin Therapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Other Study IDs: 20173CTIL
Record Dates: First submitted 2006-09-11; First posted 2006-09-12 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Non-alcoholic Fatty Liver Disease (NAFLD)
Keywords: fatty liver; statin; non-alcoholic
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver

INTERVENTIONS:
Procedure: Ultrasound to demonstrate existence of fatty liver

SUMMARY:
Aim:

1. To determine the prevalence of fatty liver in a cohort of patients hospitalized with chest pain in the Cardiology department.
2. To assess the effect of statins on the prevalence of fatty liver by a cross sectional survey of patients hospitalized with chest pain.

DETAILED DESCRIPTION:
Consecutive patients hospitalized with chest pain will be recruited at the cardiology department. Patients with an inflammatory condition, recent infection or history of alcoholism will be excluded. After signing an informed consent each patient will undergo an ultrasound examination for diagnosis of fatty liver. Information regarding BMI, hypertension and use of medications will be collected on each patient. Blood samples for fasting glucose, hemoglobin A1C, lipid profile, ESR, and CRP and liver function tests will be collected from each participant. Prevalence of fatty liver in patients who have been taking statins for 6 months or more statins will be compared to patients who have been taking statins for a lesser period and to those who do have not taken statins using a multivariate regression analysis.

Serum samples will be frozen and kept for future ongoing research.

ELIGIBILITY:
Inclusion Criteria:

* Cardiology patient
* Age above 18

Exclusion Criteria:

* Age below 18

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-09; Study Completion 2009-09 (Estimated)

REFERENCES:
- [Background] Antonopoulos S, Mikros S, Mylonopoulou M, Kokkoris S, Giannoulis G. Rosuvastatin as a novel treatment of non-alcoholic fatty liver disease in hyperlipidemic patients. Atherosclerosis. 2006 Jan;184(1):233-4. doi: 10.1016/j.atherosclerosis.2005.08.021. Epub 2005 Oct 5. No abstract available. PMID 16168995